CLINICAL TRIAL: NCT02102490
Title: A Phase 2 Study of LY2835219 for Patients With Previously Treated Hormone Receptor Positive, HER2 Negative Metastatic Breast Cancer
Brief Title: A Study of Abemaciclib (LY2835219) In Participants With Previously Treated Breast Cancer That Has Spread
Acronym: MONARCH 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15419; I3Y-MC-JPBN (Other: Eli Lilly and Company); 2013-005548-27 (Other: EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Endocrine Therapy, Taxane, MONARCH 1
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abemaciclib (Experimental): 200 milligrams (mg) abemaciclib given orally once every 12 hours for 28 days (1 cycle). Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219

SUMMARY:
The main purpose of this study is to evaluate whether the study drug known as abemaciclib is effective in treating participants with breast cancer who have already tried other drug treatments.

ELIGIBILITY:
Inclusion Criteria.

* Have a diagnosis of Hormone Receptor Positive (HR+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) breast cancer.
* Recurrent, locally advanced, unresectable or metastatic breast cancer with disease progression following anti-estrogen therapy.
* Prior treatment with at least 2 chemotherapy regimens:

  * At least 1 of these regimens must have been administered in the metastatic setting.
  * At least 1 of these regimens must have contained a taxane.
  * No more than 2 prior chemotherapy regimens in the metastatic setting.
* Have a performance status (PS) of 0 to 1 on the Eastern Cooperative Oncology Group scale.
* Have discontinued all previous therapies for cancer.
* Have the presence of measureable disease as defined by Response Evaluation Criteria in Solid Tumors Version 1.1.

Exclusion Criteria:

* Have either a history of central nervous system (CNS) metastasis or evidence of CNS metastasis on the magnetic resonance image of brain obtained at baseline.
* Received prior therapy with another cyclin-dependent kinases 4 and 6 (CDK4/6) inhibitor.
* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug.
* Have had major surgery within 14 days of the initial dose of study drug.
* Have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (27):
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - HOPE Hematology Oncology Physicians and Extenders, Tucson, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Univ of California San Francisco, San Francisco, California
  - Sansum Medical Research Foundation, Santa Barbara, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology/Hematology PA, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Presbyterian Hospital Dallas, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Texas Oncology-Sherman, Sherman, Texas
  - US Oncology, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Northwest Cancer Specialists PC, Vancouver, Washington
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleroi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Dickler MN, Tolaney SM, Rugo HS, Cortes J, Dieras V, Patt D, Wildiers H, Hudis CA, O'Shaughnessy J, Zamora E, Yardley DA, Frenzel M, Koustenis A, Baselga J. MONARCH 1, A Phase II Study of Abemaciclib, a CDK4 and CDK6 Inhibitor, as a Single Agent, in Patients with Refractory HR+/HER2- Metastatic Breast Cancer. Clin Cancer Res. 2017 Sep 1;23(17):5218-5224. doi: 10.1158/1078-0432.CCR-17-0754. Epub 2017 May 22. PMID 28533223

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Participant Flow, participants who completed were those who died due to any cause or were alive and on study at conclusion but off treatment.
Groups:
- Abemaciclib: 200 mg abemaciclib given orally once every 12 hours for 28 days (1 cycle). Participants may continue to receive treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Abemaciclib
Started | 132
Received at Least 1 Dose of Study Drug | 132
Completed | 125
Not Completed | 7
Not completed — Death | 6
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.13 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 112
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 112
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 28
  United States | 70
  France | 11
  Spain | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 14 Months)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Percentage of participants | 19.7 [13.3 to 27.5]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from first dose date to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Time Frame: From Date of First Dose until Death Due to Any Cause (Up To 27 Months)
Population: All enrolled participants who received at least one dose of study drug. Censored participants: Abemaciclib=70.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Months | 22.32 [17.72 to NA] — The upper limit of the 95% confidence interval (CI) was not calculated due to the high censoring rate.

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date.
Time Frame: From Date of CR, PR until Disease Progression or Death Due to Any Cause (Up To 14 Months)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Months | 8.6 [5.8 to 10.2]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time from the first day of therapy to the first evidence of disease progression as defined by RECIST v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 27 Months)
Population: All enrolled participants who received at least one dose of study drug. Censored participants: Abemaciclib=35.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Months | 6.0 [4.2 to 7.5]

5. Secondary Outcome: Percentage of Participants With CR, PR or SD (Disease Control Rate [DCR])
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 14 Months)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Percentage of participants | 67.4 [58.7 to 75.3]

6. Secondary Outcome: Percentage of Participants With Tumor Response of Stable Disease (SD) for at Least 6 Months, Partial Response (PR) or Complete Response (CR) (Clinical Benefit Rate)
Description: Clinical benefit rate defined as percentage of patients with best overall response of CR, PR, or SD with a duration of at least 6 months. CR, PR, or SD were defined using RECIST, v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. Percentage of participants = (participants with CR+PR+SD with a duration of at least 6 months /number of participants enrolled) *100.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 14 Months)
Population: All enrolled participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Percentage of participants | 42.4 [33.9 to 51.3]

7. Secondary Outcome: Number of Participants With Categorical Change From Baseline in Brief Pain Inventory Short Form (mBPI-sf) - Worst Pain Score
Description: A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Cycle 6 Day 1
Population: All randomized participants with a baseline and at least 1 post-baseline mBPI-sf data.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 59
Participants
  Better | 18
  No Change | 21
  Worse | 20

8. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) for Abemaciclib and Metabolites M2 and M20
Description: Area Under the Concentration versus Time Curve from Time Zero to Infinity (AUC[0-∞]) was evaluated for Abemaciclib and Metabolites M2 and M20
Time Frame: Cycle 1 Day 1 pre dose, Cycle 1 Day 15 4 hours (h) and 7 h post dose, Cycle 2 Day 1 pre dose and 3 h post dose, Cycle 3 Day1 pre dose
Population: All enrolled participants who received at least one dose of study drug (Abemaciclib) with evaluable Abemaciclib, M2 and M20 pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour/milliliters (ng*h/mL)]
Arm/Group | Abemaciclib
Number analyzed (Participants) | 132
Nanograms*hour/milliliters (ng*h/mL)]
  Abemaciclib | 3510 (38.0)
  M2 | 1620 (55.0)
  M20 | 2750 (55.0)

9. Secondary Outcome: Number of Participants With Categorical Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) - Global Health Status Score
Description: EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, cognitive, emotional, and social), global health status, and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, higher scores represent a better level of functioning. For symptoms scales, higher scores represented a greater degree of symptoms.
Time Frame: Cycle 6 Day 1
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EORTC QLQ-C30 data.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 59
Participants
  Better | 17
  No Change | 16
  Worse | 26

ADVERSE EVENTS:
Time Frame: Up To 45.57 Months
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | Abemaciclib
Serious Adverse Events (participants affected / at risk) | 33/132
Other Adverse Events (participants affected / at risk) | 132/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=132)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (2)
Cellulitis (Infections and infestations) | 2 (5)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 3 (4)
Electrocardiogram abnormal (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Renal function test abnormal (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=132)
Anaemia (Blood and lymphatic system disorders) | 35 (96)
Neutropenia (Blood and lymphatic system disorders) | 24 (88)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (21)
Lacrimation increased (Eye disorders) | 11 (12)
Abdominal pain (Gastrointestinal disorders) | 34 (54)
Abdominal pain upper (Gastrointestinal disorders) | 16 (19)
Constipation (Gastrointestinal disorders) | 27 (33)
Diarrhoea (Gastrointestinal disorders) | 120 (370)
Dry mouth (Gastrointestinal disorders) | 18 (18)
Dyspepsia (Gastrointestinal disorders) | 14 (16)
Flatulence (Gastrointestinal disorders) | 9 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (13)
Nausea (Gastrointestinal disorders) | 89 (141)
Stomatitis (Gastrointestinal disorders) | 12 (17)
Vomiting (Gastrointestinal disorders) | 46 (91)
Asthenia (General disorders) | 31 (85)
Chills (General disorders) | 8 (8)
Fatigue (General disorders) | 63 (129)
Oedema peripheral (General disorders) | 14 (16)
Pain (General disorders) | 13 (19)
Pyrexia (General disorders) | 14 (17)
Upper respiratory tract infection (Infections and infestations) | 9 (13)
Urinary tract infection (Infections and infestations) | 9 (9)
Alanine aminotransferase increased (Investigations) | 11 (15)
Aspartate aminotransferase increased (Investigations) | 12 (16)
Blood creatinine increased (Investigations) | 15 (41)
Neutrophil count decreased (Investigations) | 31 (105)
Platelet count decreased (Investigations) | 18 (42)
Weight decreased (Investigations) | 18 (22)
White blood cell count decreased (Investigations) | 24 (69)
Decreased appetite (Metabolism and nutrition disorders) | 60 (76)
Dehydration (Metabolism and nutrition disorders) | 11 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Dizziness (Nervous system disorders) | 16 (18)
Dysgeusia (Nervous system disorders) | 18 (19)
Headache (Nervous system disorders) | 26 (40)
Anxiety (Psychiatric disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (42)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days